CLINICAL TRIAL: NCT00965172
Title: A Phase II Study to Evaluate the Preliminary Efficacy Assessment of Caphosol in Patients With Sarcoma Receiving Multicycle Chemotherapy With Doxorubicin and Ifosfamide or Cisplatin
Brief Title: Caphosol in Sarcoma Patients With Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0276
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Sarcoma; Oral Mucositis
Keywords: Cancer; Mucositis; Chemotherapy; Caphosol; Calcium phosphate; Sodium Bicarbonate; Baking Soda Solution; Multi-cycle chemotherapy
MeSH Terms: conditions — Sarcoma; Stomatitis; Neoplasms; Mucositis | interventions — calcium phosphate; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caphosol (Experimental): Caphosol (calcium phosphate)
  Interventions: Other: Caphosol
- Baking Soda (Active Comparator): Control Group (standard of care)
  Interventions: Other: Baking Soda

INTERVENTIONS:
Other: Caphosol — Oral rinse of calcium phosphate solution five times daily beginning on day one of chemotherapy.
  Other Names: calcium phosphate
  Arms: Caphosol
Other: Baking Soda — Oral rinse of baking soda solution as per standard of care five times daily beginning on day one of chemotherapy.
  Other Names: Sodium Bicarbonate
  Arms: Baking Soda

SUMMARY:
The goal of this clinical research study is to find out if Caphosol® (calcium phosphate) mouthwash is more effective than a baking soda solution at preventing and treating mucositis, in patients with sarcoma who are to be treated with chemotherapy. The safety of this drug will also be studied. Researchers also want to learn about the way calcium phosphate may affect mucous membranes.

The goal of this clinical research study is to see if Caphosol® (calcium phosphate) mouthwash is better than baking soda solution in patients with sarcoma who are to be treated with chemotherapy . Caphosol will also be studied to see if it lessens the incidence and severity of oral mucositis (painful sores in the mouth).

DETAILED DESCRIPTION:
Chemotherapy and radiation therapy can hurt normal cells in the gastrointestinal tract (which includes the mouth and intestines). When this happens, it can cause mucositis (inflammation of the lining of the mouth, throat, and intestines). Researchers want to compare the effects of calcium phosphate and baking soda on patients who are at risk for mucositis.

The Study Drugs:

Caphosol (calcium phosphate) is a saliva-like liquid that is designed to replace the chemical and pH (acid) balance in the mouth. It is used as a mouth rinse to moisten, lubricate, and clean the mouth, including the lining of the mouth, tongue, and throat. It is also used to loosen thick mucous and help prevent the mucous membranes from sticking together.

Baking soda is used as the standard of care for preventing and treating mucositis.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to receive either calcium phosphate mouth rinse or the baking soda mouth rinse during the study. There is an equal chance of being assigned to either group.

You will use the mouth rinse 5 times every day. The study staff will explain how to mix and rinse with it.

Calcium phosphate should be stored at room temperature and should not be refrigerated. If you are on a low sodium diet, you should check with your doctor before using calcium phosphate.

Baseline Tests:

The following tests and procedures will be performed before you receive your first dose of chemotherapy:

* Blood (about 3 teaspoons) will be drawn for routine tests.
* The mucous membranes in your mouth will be checked.
* You will be asked to complete a questionnaire (about 15 minutes) on how you feel.
* You will be given a diary before you start each cycle to record if you have any mouth pain.

Study Tests:

You will need to come to MD Anderson on around Days 10, 12, and 14 (depending on the status of the mucositis) of each chemotherapy cycle. During these clinic visits, the following tests and procedures may be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* The mucous membranes in your mouth will be checked. Also, you may have your mouth and throat photographed.
* You will be asked to complete the questionnaire on how you feel.
* When possible, the optical imaging procedures will also be performed on these days.

Length of Study and Reasons for Leaving the Study Early:

You will take part in this study for up to 18 weeks (4 to 5 months). You will be taken off study if you experience intolerable side effects.

End of Study Visit:

You will also have an end of study visit after you complete 6 cycles of study drug, if you are taken off study for any reason, or if you choose to leave the study. During this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* The mucous membranes in your mouth will be checked.
* You will be asked to complete the questionnaire on how you feel.
* You will receive a phone call from the nurse after you last dose of study drug to follow up on any side effects.

This is an investigational study. Caphosol (calcium phosphate) is FDA approved and commercially available for use in preventing and treating mucositis, and for relief of dry mouth during high dose chemotherapy or radiation treatment.

Up to 30 patients will take part in this study. All will be enrolled at M. D Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoma which is locally advanced, at high risk for relapse or metastatic for whom treatment with high dose doxorubicin (75-90 mg/m^2) with ifosfamide (AI) or cisplatin (AP) is indicated.
2. Must be >16 and < 65 years of age.
3. Females of childbearing potential (defined as not post-menopausal for 12 months, or no previous surgical sterilization) must have a negative blood pregnancy test.
4. Male and Females of child bearing potential must use acceptable methods of birth control which include oral contraceptives, spermicide with either a condom, diaphragm or cervical cap, us of a intrauterine device (IUD) or abstinence.
5. Adequate hematologic (ANC > 1500/mm^3, platelet count > 150,000/mm^3), renal (serum creatinine < 1.5mg/dL), hepatic (serum bilirubin count < 1.5 x normal and SGPT <3 x normal) functions.
6. Karnofsky Performance Status >/= 80%
7. Signed informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with any co-morbid condition which renders patients at high risk of treatment complication.
3. Patient has uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%), uncontrolled cardiac arrhythmia or hypertension, acute myocardial infarction within 3 months
4. Patient has an active seizure disorder. (Patients with a previous history of seizure disorders will be eligible for the study, if they have had no evidence of seizure activity, and they have been free of antiseizure medication for the previous 5 years.)
5. Prior surgery or radiotherapy (RT) within 2 weeks of study entry.
6. Psychological, social, familial, or geographical reasons that would prevent scheduled visits and follow-up.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence/Severity of Oral Mucositis WHO Grades 1, 2, 3, and 4 | Incidence of mucositis (all grades) within 6 cycles of treatment (estimate 18 weeks, 4 to 5 months).

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org